CLINICAL TRIAL: NCT06112431
Title: Eye Health Intervention Study in Upper Manhattan
Acronym: EYES-UM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Lisa Hark, PhD, MBA, Professor of Ophthalmic Sciences, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: AAAV6542; PA-25-305 (Other Grant/Funding Number: National Eye Institute)
Record Dates: First submitted 2023-10-26; First posted 2023-11-01 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Glaucoma, Suspect; Diabetic Retinopathy; Cataract; Refractive Errors; Vision Impairment and Blindness
Keywords: Randomized Clinical Trial; Implementation Outcomes; Eye Health Intervention; Glaucoma/Glaucoma Suspect; Eye Health Screenings and Optometric Exams; Leading Causes of Eye Disease; Telehealth Image Reading; Vision Health Policy Roadmap
MeSH Terms: conditions — Ocular Hypertension; Diabetic Retinopathy; Cataract; Refractive Errors; Vision Disorders; Blindness | interventions — Methods

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Ophthalmologists reading the fundus images will be masked to randomization assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Participants randomized to the Intervention Arm and referred to ophthalmology will receive assistance from a Study Coordinator with scheduling in-office eye exam appointment and arranging transportation to these appointments over 2 years at either Columbia Ophthalmology, Harlem Hospital, or their own eye care provider.
  Interventions: Other: Intervention
- Usual Care (Placebo Comparator): Consented participants randomized to the Usual Care Arm will receive all the basic level of services including the eye health screening, optometric exam if they fail the screening, and eyeglasses at no charge. Those who require referral to ophthalmology will be scheduled for the initial in-office eye exam and their outcomes will be tracked. No additional support will be provided the Usual Care participants during the study. The Usual Care Arm represents a realistic choice currently available for participants following eye health screening.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Intervention — Participants randomized to the Intervention Arm and referred to ophthalmology will receive assistance from a Study Coordinator with scheduling in-office eye exam appointment and arranging transportation to these appointments over 2 years at either Columbia Ophthalmology, Harlem Hospital, or their own eye care provider.
  Arms: Intervention Arm
Other: Usual Care — Consented participants randomized to the Usual Care Arm will receive all the basic level of services including the eye health screening, optometric exam if they fail the screening, and eyeglasses at no charge. Those who require referral to ophthalmology will be scheduled for the initial in-office eye exam and their outcomes will be tracked. No additional support will be provided the Usual Care participants during the study. The Usual Care Arm represents a realistic choice currently available for participants following eye health screening.
  Arms: Usual Care

SUMMARY:
Individuals living in Upper Manhattan have limited access to eye care, high vision impairment rates, and poor ocular health outcomes. To improve eye care and vision health outcomes, the Eye Health Intervention Study in Upper Manhattan (EYES-UM) will conduct eye health screenings in accessible primary care health centers and senior centers and implement a behavioral intervention to improve adherence for those referred for in-office eye care. The proposed innovative, 2:1 cluster-randomized clinical trial, will recruit adults age 40 and older in Upper Manhattan with known rates of inadequate eye care. A total of 10 settings in Upper Manhattan, comprised of primary care offices, senior centers, and organizations, confirms access to 17,000 individuals living at or below the NYC.gov poverty measure. This study will conduct ocular tests (visual acuity, intraocular pressure, fundus images) during screenings. To ensure that all participants receive the basic level of service, all participants who fail the eye health screening will be seen the same day by a study optometrist and eyeglasses will be provided at no charge. Educational workshops and an Advisory Board will support recruitment. Intervention Arm participants will receive ongoing support with scheduling eye exams and transportation by trained Study Coordinators. All participants will be followed prospectively for 2 years. The study is guided by the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) Framework. Conducting Focus Groups with health policy stakeholders ensures iterative input during the study to bridge and translate EYES-UM findings into a Vision Health Policy Roadmap for scalable implementation of vision care delivery models, focusing on adherence.

DETAILED DESCRIPTION:
Populations in urban settings such as Upper Manhattan, have limited access to eye care, high vision impairment rates, and poor ocular health outcomes. Our team of vision researchers designed the Eye Health Intervention Study in Upper Manhattan (EYES-UM) to provide eye health screenings directly in Upper Manhattan, in familiar and accessible settings. The proposed innovative, 2:1 cluster-randomized clinical trial, will recruit adults age 40 and older in Upper Manhattan with high rates of inadequate eye care.

A total of 10 settings in Upper Manhattan, comprised of health centers and senior centers, confirms access to 17,000 individuals. This study will conduct ocular tests (visual acuity, intraocular pressure, fundus images) during screenings. To ensure that all participants receive the basic level of service, all participants who fail the eye health screening will be seen the same day by a study optometrist and eyeglasses will be provided at no charge. Educational workshops and an Advisory Board will support recruitment. Intervention Arm participants will receive ongoing support with scheduling eye exams and transportation by trained study coordinators. All participants will be followed prospectively for 2 years. The study is guided by the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) Framework: In Aim 1, we will evaluate the effectiveness of an Eye Health Intervention to improve access to vision health services in 10 settings in Upper Manhattan. After eye health screenings and optometric exams, we will conduct a 2:1 cluster-randomized clinical trial using an Intervention to provide eye exam scheduling and transportation for those referred to ophthalmology to improve in-office eye exam adherence behavior over 2 years (primary implementation outcome) and eye disease detection (primary clinical effectiveness outcome). In Aim 2, using the RE-AIM Framework, we will evaluate the implementation of the Eye Health Intervention using mixed-methods. Aim 3 includes a proactive implementation science approach to produce a real-world Vision Health Policy Roadmap by conducting Focus Groups with health policy stakeholders to understand evidence needed to develop scalable and sustainable nationwide vision care delivery models and how to incentivize payors to ensure the success of these efforts. The Eye Health Intervention will protect and improve vision health outcomes and provide a sustainable model that can be scaled-up in many settings. By providing basic eye care services and eyeglasses to all participants, simplifying access and supporting utilization of in-office eye care, this innovative research strategy will generate important evidence and a roadmap for policy change to advance vision health. This innovative approach using Focus Groups ensures iterative input during the study to bridge and translate EYES-UM findings into a Vision Health Policy Roadmap for scalable implementation of vision care delivery models, focusing on adherence.

ELIGIBILITY:
Inclusion Criteria:

* Individuals age 40 years or older.
* Living independently.

Exclusion Criteria:

* Self-reported terminal illness with life expectancy of less than 1 year.
* Inability to provide informed consent due to dementia or other reason.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5840 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2031-03-31 (Estimated); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
Primary Implementation Outcome: Adherence to IN-OFFICE Eye Exam for those referred to ophthalmology | 2 years
  The primary implementation outcome measure for Aim 1 is ADHERENCE TO IN-OFFICE eye exam for those referred to ophthalmology and will be measured by appointment attendance at the initial in-office eye exam appointment for those referred to ophthalmology. The unit of measure is the eye exam appointment, which will be scheduled within 6-months (+/-4 months) of the referral at either Columbia Ophthalmology, Harlem Hospital or their own eye care provider. The measure will assess the rate of adherence at the initial appointment. Comparisons will be made between the Intervention Arm and the Usual Care Arm.
Primary Clinical Effectiveness Outcome: Detection of Eye Disease | 2 years
  The primary clinical effectiveness outcome measure for Aim 1 is detection of eye disease(s) (glaucoma, retina, other) confirmed by in-office eye exams and will be measured by rates of detection of eye disease(s) for those referred to ophthalmology. All initial in-office eye exams will be scheduled at the conclusion of eye health screenings. Outcome measures will assess rates of eye disease detection, specifically glaucoma/suspect, among those referred to ophthalmology. A comparison will be made between participants living in the 7 health settings randomized to the Intervention Arm compared to 3 settings randomized to Usual Care Arm. Participants who request their own eye doctor, the medical release form will be signed, and we will schedule the eye exam, so we can also track attendance.

SECONDARY OUTCOMES:
Return Attendance at Eye Health Screenings at 1, 2, and 3 Years | 1, 2, and 3 years
  As a safety net, all participants will be informed of the future dates of the eye health screenings but not required to attend. We hypothesize that participants will return at various intervals (1, 2, and/or 3 times) and we want to understand the demographic and clinical characteristics of these participants as well as the frequency of attendance and why they returned and compare to those who do not participate again at the health setting. The intervals will be 12, 24 or 36 months and we will measure the number and percentage of participants who attend the eye health screenings over 4 years. We will provide descriptive statistics of participants who re turn to the eye health screenings at these intervals to understand the characteristics associated with return attendance.
Follow-up Adherence to Recommended In-office Eye Exams at 1 - 4 Years | 4 years
  A maintenance measure is adherence to recommended in-office eye exams for those who attend the initial eye exam to determine access to care sustainability and will be reported by randomization group. Adherence will be assessed annually on the basis of the expected follow-up schedule defined at the index visit for that year if the participant attends. In the first year, the follow-up recommendation given by the ophthalmologist will be classified into 1 of 4 categories: return within 2 months, return in 3 to 4 months, return in 6 months, or return in 12 months. This follow-up recommendation will be translated into the corresponding expected number of visits per year: 6, 3, 2, or 1.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A. Hark, PhD, MBA, Principal Investigator — Columbia University Department of Ophthalmology
Locations (1):
- Cuimc/Nyph, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No